CLINICAL TRIAL: NCT01556347
Title: Multi-Drug Desensitization Protocol for Heart Transplant Candidates
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Timothy Icenogle, MD, Director, Inland Northwest Thoracic Transplant Program, Providence Health & Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND110875
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Heart Transplantation
Keywords: alloantibody; immunologic; memory; heart; transplant; desensitization
MeSH Terms: interventions — Bortezomib; thymoglobulin; Rituximab; Immunoglobulins, Intravenous; Plasmapheresis; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Elimination of Immunologic Memory (Experimental): A single arm multi-drug regimen is used to delete immunologic memory in order to reduce or eliminate alloreactive anti-HLA antibodies in highly sensitized heart transplant candidates. The intervention includes a protocol of Thymoglobulin, Rituximab, plasmapheresis and Bortezomib.
  Interventions: Drug: Bortezomib, Thymoglobulin, Rituximab, Gamimune N, (IVIG), Plasmapheresis

INTERVENTIONS:
Drug: Bortezomib, Thymoglobulin, Rituximab, Gamimune N, (IVIG), Plasmapheresis
  Other Names: Anti-thymocyte globulin (rabbit), Rituxan, Velcade

SUMMARY:
Background: Patients may develop antibodies (human leukocyte antigen [HLA] alloantibodies) to other human tissues via pregnancy, transfusions or previous transplantation, which limits the ability to find an acceptable donor heart for transplantation. Such patients are at high risk for antibody mediated rejection, graft failure, and acute rejection (i.e. death). For successful transplantation, patients must receive organs from donors who lack the HLA antigens that correspond to their alloantibody specificities. No successful desensitization strategy currently exists.

Purpose: To determine if desensitization by deletion of immunologic memory with a multi-drug approach including anti-T and B cell therapies and anti-plasma cell therapy can effectively eliminate or significantly reduce alloantibody levels and permit highly sensitized patients to obtain a heart transplant. This therapy is anticipated to remove immunologic memory and will require re-immunization.

DETAILED DESCRIPTION:
Transplant candidates with HLA alloantibodies are at high risk for antibody mediated rejection (AMR), graft failure, and acute rejection (1,2). In heart transplantation, these complications lead to death. The 50% calculated panel reactive antibody, CPRA, threshold is chosen from a consensus statement from the International Society of Heart and Lung Transplantation (3). This value is admittedly arbitrary but does represent a consensus of accepted opinion amongst experienced and reputable heart transplant centers.

The alloantibodies that prevent these patients from being transplanted are a result of the adaptive immune system and immunologic memory. Immunologic memory is defined as the ability of the immune system to provide a faster, stronger and more specific response to a second exposure of an antigen, when the antigen was completely eliminated from the organism after the prior exposure.

There are three major cell lines involved in immunologic memory: memory T cells, memory B cells and plasma cells, all of which can survive once antigen has been eliminated (4). B cells can mount responses to both small soluble antigens and large antigens (5). Once a B cell becomes activated, it can become a short lived plasma cell and produce immunoglobulin M, (IgM), antibodies or it can enter a germinal center where it can undergo somatic hypermutation with affinity maturation and isotype switching. The B cell can then differentiate into a long lived plasma cell and compete for a bone marrow niche or can become a memory B cell (4-8).

Memory T cells can last a lifetime and can recirculate between the secondary lymphoid organs (SLO) as central memory T cells (TCM) or in the peripheral tissues as effector memory T cells (TEM) (4,9). Upon encountering their cognate antigen, they can rapidly proliferate and differentiate to effector T cells.

Memory B cells slowly proliferate and recirculate in the SLOs, last there for decades and memory B cells to vaccinia (smallpox) have been noted to survive for more than 50 years (9). They are commonly identified by the presence of CD27 and upon a second antigenic challenge; the memory B cells can rapidly proliferate and then differentiate into new plasma cells (10). This phenomenon provides a redundant system or "array" to replenish plasma cells that produce antibody for a given antigen.

Plasma cells are highly differentiated and specific cells that can actively produce alloantibody. There are two populations of plasma cells, short-lived and long-lived (8). Long-lived plasma cells can last for life and can appear within less than 1 week of antigenic stimulation (6,7). In core biopsies of kidney transplant recipients, B cells, memory B cells, plasmablasts and plasma cells have all been identified during acute rejections (11). The plasma cells are end differentiated and therefore cannot proliferate. In the bone marrow, there are a finite number of survival niches (109) dependent on the number of stromal cells present to support them. Plasma cells that don't find sanctuary in the marrow or lose sanctuary only last a few days, probably owing to the intense metabolic demands of a cell that can produce between 10,000 to 20,000 copies of antibody per second (12). Plasma cells are currently thought as being without a negative feedback loop to suppress their antibody synthesis. Plasma cells have been demonstrated to have an FcγRIIB receptor coupled to an immunoreceptor tyrosine based inhibitory motif (ITIM) (13). The FcγRIIB receptor is a low affinity receptor and cannot bind monomeric immunoglobulin G, (IgG). The homeostasis of immunoglobulin is thought to be mainly the responsibility of the endothelial cell (14). Once an antibody is produced, endothelial cells can eliminate circulating antibody by lysosomal degradation or recycling the antibody through an Fc receptor neonatal, (FcRn) dependent mechanism back into the plasma.

A successful plan to eliminate the memory of a given antigenic encounter must address the three separate systems or "arrays." The elimination of immunologic memory such that deleterious antibodies could be removed and then new favorable antibodies created would be a significant advance in the fields of transplantation and autoimmunity. A review of the medications used in IND 110875 will elucidate why this protocol may be successful where all others have failed.

Rabbit antithymocyte globulin, RATG, has anti-T-cell properties, and in particular, activity against memory T-cell surface antigens, thereby causing complement mediated T-cell death in peripheral blood and apoptosis in the spleen and lymph nodes (15). RATG has antibodies to CD27, CD38, HLA-DR and has demonstrated anti-memory B cell properties in vitro and in vivo (15-17). The combination of rATG and rituximab decreased CD27 positive B cells from the spleen in patients in a desensitization trial that was otherwise unsuccessful was a significant observation (16).

Rituximab, an anti-CD20 monoclonal antibody, has strong activity against B-cells and depletes B cells in the circulation for 5-7 months. But as B-cells differentiate into plasma cells, the CD20 surface marker is down regulated, with concomitant loss of sensitivity to rituximab (18). Rituximab has been used in a variety of autoimmune diseases (19,20). Many antibodies are not affected while others are decreased for a period of time. Short lived plasma cells may be decreased since there is not a ready supply of B cells to replace them after their short three day half-life. In a study in systemic lupus erythematosis (SLE) using rituximab; flow cytometry and autoantibody specificity studies revealed that antibodies to Ro52 and La44 and measles were not decreased but antibodies to dsDNA and C1q did decrease (19). The overall amount of immunoglobulin did not change. Plasma cells are not affected by anti-CD20, so the antibody production from long lived plasma cells continues unabated. Memory B-cells are CD 27+ and have a variable expression of CD20. A study in desensitizing kidney transplants candidates showed that rituximab did not decrease the number of CD27+ memory B cells or plasma cells in the spleen (16). In (SLE) patients treated with rituximab the cells returning after depletion were largely naïve B cells and the plasmablasts were 2.3 times higher than at baseline (19). While memory B cells circulating in the blood were lower after rituximab therapy, the memory B cells in the spleen appear to be unaffected and can then transform in to plasmablasts which can then secrete soluble antibody. This observation explains why some antibodies will disappear, at least temporarily with rituximab while others will not. If the antibody is coming primarily from short lived plasma cells or plasmablasts, rituximab will more likely have an effect; these antibodies are produced by cells with a short half-life and are dependent upon continuous proliferation of B cells. Antibodies produced by long-lived plasma cells are not affected by rituximab. Rituximab does not affect memory B cells in the spleen, so they can rapidly reform plasmablasts and plasma cells to reconstitute the cell lines producing certain clones of antibodies. Since memory B-cells can become antibody secreting plasma cells, it is advantageous to remove them before transplantation in the highly sensitized patient.

The combination of rATG and rituximab was shown in the human to reduce memory B cells in the spleen (16). This finding has not yet been incorporated into a desensitization protocol or into a protocol for autoimmune therapies from our review of the literature. No other therapy effectively reduces memory B cells in the human and it represents a novel aspect of IND 110875.

No agents previously used in transplantation, including rATG and rituximab, have the ability to inhibit mature plasma cells once they find refuge in the bone marrow, and therefore have little effect on reducing antibody production. However, bortezomib, a proteasome inhibitor used in treatment of multiple myeloma, does have the ability to deplete plasma cells via many mechanisms.

Proteasome inhibition represents a novel treatment strategy because it provides a means for depleting plasma cells within the bone marrow (21,22). Bortezomib is approved for use in the treatment of multiple myeloma and the sensitivity of myeloma cells to proteasome inhibitors is proportional to their immunoglobulin synthesis rates (22). Plasma cells are known to have high immunoglobulin synthesis rates and treatment with bortezomib depleted both short and long-lived plasma cells by more than 60% in the spleen and 95% in the bone marrow after 48 hours of treatment in the BALB/c mouse model. Bortezomib activated the unfolded protein response (UPR) documented by increases in the expression of the chaperones BiP and Chop which are markers for UPR. The authors also concluded that the late inhibition of the anti-apoptotic transcription factor NF-κB also contributed to cell death. In a lupus nephritis mouse model (NZB/W F1 mice) treated with bortezomib, dsDNA-specific antibodies decreased to the range of non-autoimmune mice. Total serum IgG, IgG2a, IgG3, IgM, and IgA concentrations were all strongly reduced but concentrations of IgG1 and IgG2 were not altered or only slightly altered (21). Total IgG concentrations were not reduced by more than 50%. The authors noted that newly formed plasma cells could return by 48 hours after bortezomib injection. These findings support the conclusion that bortezomib can kill plasma cells, and have a salutary clinical effect, but memory B cells are not depleted and plasma cells can quickly recover and produce unwanted antibody. The ability of bortezomib to kill non-malignant plasma cells represents a major finding with potential therapeutic efficacy in transplantation and autoimmune diseases, but by itself is incapable of long lasting reductions in antibody. The clinical finding of variable reductions in antibody levels with bortezomib can be explained from these findings in the basic science literature.

Bortezomib has been used as a rescue strategy for the treatment of refractory antibody mediated rejection (23-25). An in vitro study revealed that bortezomib was able to induce apoptosis in plasma cells aspirated from renal transplant recipients whereas rATG, rituximab and IVIG all failed to cause apoptosis (25). Treatment with bortezomib at concentrations that blocked antibody production in vitro was shown to significantly decrease the 20S proteasome chymotrypsin-like peptidase activity. Two patients had bone marrow biopsies during acute humoral rejection, one week after bortezomib and one year later which revealed that the total number of plasma cell allospecificities decreased as did the total percentage of plasma cells (25). Not all antibodies were reduced by bortezomib in these two patients and the total IgG levels were unchanged, yet this study did show that bortezomib could decrease plasma cells in the bone marrow.

Bortezomib is indicated for multiple myeloma wherein the malignant plasma cells are very aggressive in producing antibody. The more productive the myeloma cell line is to making antibody, the more susceptible to proteasome inhibition (22). The above literature in non-malignant plasma cells also reveals that they are susceptible to proteasome inhibition with bortezomib, but in a number of studies, certain immunoglobulin fractions did not decrease and the overall amounts of immunoglobulin were unchanged. Perhaps plasma cells are not as metabolically active as their malignant counterparts. There is some evidence that plasma cells may be able to decrease their immunoglobulin synthesis and this in turn would make them less susceptible to proteasomal inhibition (26). A reexamination of immunoglobulin homeostasis reveals a potential therapy to increase sensitivity to bortezomib.

Immunoglobulin homeostasis is largely felt to be the result of plasma cell production and then FcRn mediated recycling in the endothelial cells. Antibody that does not combine with FcRn in the endosome of the endothelial cell is then degraded while antibody that does combine is recycled back to the interstitial space (27). The concept that IgG does not have a negative feedback loop to the plasma cell is supported by data in the experimental animal and humans (28,29). However, clinicians observe patients that "rebound" after plasmapheresis with levels of antibody that were just as high or higher than before plasmapheresis and this led to the conclusion that there was a negative feedback loop (30,31). The rebound phenomenon was explained away as the return of antibody from the periphery and increased recycling by FcRn receptors (28). The regulation of protein synthesis in the plasma cell has received new attention and is controlled by a complex system of feedback loops involving the endoplasmic reticulum stress and mTOR signaling (32).

Recent investigations into the mechanism of intravenous immunoglobulin, IVIG, function offer further insight into possible explanation for a negative feedback loop to plasma cells. IVIG in the clinical literature is thought to work by a number of pathways including anti-idiotypic antibodies, inhibition of cytokine gene activation, anti-T cell receptor activity, anti CD4 activity, stimulation of cytokine receptor antagonists, inhibition of complement activity and Fc mediated interactions with antigen presenting cells to block T cell activation (33). Recent work reveals that these mechanisms are possibly erroneous. Studies in children with ITP in 1993 revealed that infusion of Fc fragments provided the anti-inflammatory properties (34). The anti-inflammatory properties of IVIG can now be attributed to Fc sialylation of IgG (35-37). Immunoglobulins are glycoproteins and a single N-linked glycan is found at Asn297 in the Fc domain. This covalently linked complex glycan is composed of a biantennary heptapolysaccharide containing N-acetylglucosamine and mannose and two terminal sialic acid residues (35). Further modifications of this carbohydrate structure are common and over 30 different glycans have been identified at this one site and glycosylation of IgG is mandatory for FcγR binding. The total anti-inflammatory activity of IVIG depends on the sialylation of the IgG Fc fragments and this represents only 5% of the IgG pool. The small amount of sialylated IgG in IVIG explains why large doses are required for its anti-inflammatory effects while much lower doses are required to treat hypogammaglobulinemia. Plasmapheresis, by decreasing sialylated IgG, may lead to the up-regulation of antibody synthesis in plasma cells and make them more susceptible to bortezomib.

The index patient treated with a protocol similar to this one, the patient had effective deletion (< 5000MFI) of all of their antibodies detected by LABScreen, including the Class II antibodies that prior to this had been difficult to remove. Using the much more stringent criteria of < 1000 MFI, the index patient had only one remaining antibody over 1000 at the end of 3 cycles of the bortezomib treatment phase. The patient was unique amongst the case reports of therapies for antibody mediated rejection and desensitization therapy in that all of the patient's antibodies dramatically declined and the total amount of soluble antibody decreased to the point where the patient required IVIG for replacement therapy. If this result is reproducible and the protocol has sufficient safety, then these results could have important ramifications in the fields of transplantation and autoimmune disease. Autoantibody mediated diseases may now have the potential of cure if the immunologic memory of the inciting epitopes is erased.

It is impossible to study these medications in the usual one-drug-at-a-time methodology given the redundant nature of immunologic memory. The potential risk of the protocol is only acceptable because of the need to develop an effective therapy for a life-threatening situation. This protocol is in line with the criteria elucidated by the FDA in the recent New England Journal of Medicine article, "Development of Novel Combination Therapies" (38). The article mainly describes combination therapies for cancer trials; however, the thematic components of the document apply to IND 110875.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary signed informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

  2.Female subject is either post-menopausal or surgically sterilized, or willing to use two acceptable methods of birth control for the duration of the study and for up to 2 months after the last dose of study medication.

  3.Male subject agrees to use an acceptable method for contraception for the duration of the study.

  4.Patient is greater than or equal to 18 years of age but less than 70 years old (inclusive).

  5.Patients with a Calculated Panel Reactive Antibody (CPRA) of ≥ 50% by Luminex Single Antigen Flow Bead (SAFB) testing (LABScreen®, Canoga Park, CA), where a Mean Fluorescence Intensity (MFI) of 1000 is the positive threshold.

  6.Patient is considered compliant and intends to be available for follow-up study period of 1 year.

  7.Patient must have no known hypersensitivity to treatment with bortezomib, boron, or mannitol.

  8.Patient must have no hypersensitivity to rituximab. 9.Patient must have no history of allergy or anaphylaxis to rabbit proteins or to any product excipients, or have active acute or chronic infections which contraindicate additional immunosuppression.

  10.Patient must have no history of an anaphylactic or severe systemic response to Immune Globulin (Human). Individuals with selective IgA deficiencies who have antibody against IgA (anti-IgA antibody) should not receive IVIG since these patients may experience severe reactions to the IgA which may be present.

  11.Patients without an AICD implanted will need to consent to wear a Zoll LifeVest Wearable Defibrillator.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or have a positive pregnancy test on enrollment. If the patient becomes pregnant during the study, she must be removed from the study before receiving any additional study drug.
2. History of hepatitis C virus (HCV) positivity (by polymerase chain reaction, PCR)
3. Patients who are human immunodeficiency virus (HIV)-positive, or hepatitis B surface antigen (HBsAg)-positive.
4. Patient is deemed likely to have a second solid organ transplant or cell transplant (e.g. kidney or islet cell) in next 3 years.
5. Patient at risk for tuberculosis (TB):

   1. Current clinical, radiographic, or laboratory evidence of active or latent TB as determined by local standard of care
   2. History of active TB:
   3. Within the last 2 years, even if treated
   4. Greater than 2 years ago, unless there is documentation of adequate treatment according to locally accepted clinical practice
   5. Patient at risk of reactivation of TB precludes administration of conventional immunosuppression (as determined by investigator and based upon appropriate evaluation)
6. Patient with active peptic ulcer disease (PUD), chronic diarrhea, or gastrointestinal malabsorption
7. Patient with a history of hypercoaguable state
8. Patient with hemoglobin < 7 g/dL, white blood cell (WBC) count < 2000/mm3 (3 x 109/L) or platelet count < 30,000 /mm3 prior to transplant
9. Receipt of a live vaccine within 4 weeks prior to study entry
10. Patient treated with immunosuppressive therapy (e.g. methotrexate, abatacept, etc) for indications such as autoimmune disease, or patient with comorbidity to a degree that treatment with such agents is likely during the trial in the opinion of the investigator
11. Patients with current or recent severe systemic infections within 2 weeks of medication start
12. Evidence of severe liver disease with abnormal liver profile (aspartate aminotransferase [AST], alanine aminotransferase [ALT] or total bilirubin > 1.5 times upper limit of normal (ULN) at screening.)
13. Patient has ≥ Grade 2 peripheral neuropathy within 14 days of medication start
14. History of malignancy within the past 5 years that is not considered to be cured, with the exception of localized basal cell carcinoma of the skin (excised ≥ 2 years prior to study initiation)
15. Prisoner or patient compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g. infectious disease) illness
16. Patient with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not compatible with adequate study follow-up
17. Patient with a history of amiodarone exposure within three months.
18. Patient with a previous heart or other transplant

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiimothy B Icenogle, MD, Principal Investigator — Providence Sacred Heart Medical Center
Locations (1):
- Providence Sacred Heart Medical Center, Spokane, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The candidates for this study were recruited from the clinic of the Inland Northwest Heart Transplant and Mechanical Heart Program at Providence Sacred Heart Medical Center in Spokane, Washington. The Study received final IRB approval Jan. 4, 2013 after having received FDA approval.
Pre-assignment Details: The potential candidates had to be accepted heart transplant candidates who met a stringent list of inclusion and exclusion criteria to become study candidates.
Groups:
- Highly Sensitized Heart Transplant Candidates: This was a Single Group Assignment Interventional Study to determine if a multi-drug regimen could be used to delete immunologic memory in order to reduce or eliminate alloreactive anti-HLA antibodies in highly sensitized heart transplant candidates. It was a non-randomized, open label, safety/efficacy (pilot) treatment study. It was hoped that if the calculated panel reactivity antibody (CPRA) was reduced to less than 20% via the protocol, then the patients could become functionally transplantable. There were three phases of the study, an Induction Immunotherapy Phase, a Bortezomib Treatment Phase, and a Recovery Phase. Both patients completed each of the three phases.
Period: Induction Immunotherapy
Arm/Group | Highly Sensitized Heart Transplant Candidates
Started | 2
Completed | 2
Not Completed | 0
Period: Bortezomib Treatment Phase
Arm/Group | Highly Sensitized Heart Transplant Candidates
Started | 2
Completed | 2
Not Completed | 0
Period: Recovery Phase
Arm/Group | Highly Sensitized Heart Transplant Candidates
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Heart transplant candidates with a CPRA greater than 50% who underwent a multi-drug therapy to eliminate immunological memory.
Groups:
- Elimination of Immunologic Memory: A Multi-drug regimen is used to delete immunologic memory in order to reduce or eliminate alloreactive anti-HLA antibodies in highly sensitized heart transplant candidates.
  Bortezomib, Thymoglobulin, (rATG), Rituximab, Gamimune N, (IVIG), Plasmapheresis (Multidrug Protocol): Bortezomib, Thymoglobulin, (rATG), Rituximab, Gamimune N, (IVIG), Plasmapheresis
Arm/Group | Elimination of Immunologic Memory
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants] — Heart transplant candidates with CPRA > 50%
  Participants
    United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Reduction in CPRA to Less Than 20%
Description: Percentage of highly sensitized heart transplant candidates, (patients with a CPRA greater than 50%), who have desensitization therapy, and then achieve a reduction in alloantibody such that their CPRA falls below 20%. For an individual patient, the outcome measure time frame is the one year of the Recovery Phase which begins after 218 days from the time that the patient begins the Induction Immunotherapy Phase, which is the same as the end of the Bortezomib Treatment Phase.
Time Frame: 365 days
Population: There were two patients entered into the study and therefore two patients analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Highly Sensitized Heart Transplant Candidates: The percentage of patients with a CPRA less than 20% during the Recovery Phase of the protocol
Arm/Group | Highly Sensitized Heart Transplant Candidates
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Percentage of Patients Transplanted
Description: Percentage of patients, who are transplanted within one year of finishing the Bortezomib treatment phase.
Time Frame: 365 days
Population: The two patients who were entered into the study were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Highly Sensitized Heart Transplant Candidates: Highly sensitized heart transplant candidates with a CPRA greater than 50% that complete the Bortezomib treatment phase and are transplanted within one year
Arm/Group | Highly Sensitized Heart Transplant Candidates
Number analyzed (Participants) | 2
Participants | 0

3. Primary Outcome: Percentage of Patients Who Suffer Mortality, a Serious Adverse Event, or Other Adverse Event During the Study Period
Description: Percentage of study patients who experience a serious safety issue during the three phases of the study as measured by all cause mortality, serious adverse reactions and other adverse reactions.
Time Frame: 583 days
Population: Two patients were entered into the study and both were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- All Cause Mortality: Mortality for any reason during the study period
- Serious Adverse Events: The number of study patients with serious adverse events.
- Other Adverse Events: The number of study patients who had adverse events other than serious.
Arm/Group | All Cause Mortality | Serious Adverse Events | Other Adverse Events
Number analyzed (Participants) | 2 | 2 | 2
Participants | 0 | 2 | 2

4. Primary Outcome: Percentage of Patients Who Experience Grade 3 and Above Non-Hematologic Toxicities
Description: Percentage of patients who experience of grade 3 and above non-hematologic toxicities as measured by the incidence of hypersensitivity reaction, fever, nausea and vomiting or dehydration during the study period.
Time Frame: 583 days
Population: There were two patients entered into the study and both were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Patients With Grade and Above Non-Hematologic Ti: Percentage of patients who experienced a Grade 3 or above non-hematologic toxicity during any phase of the study
Arm/Group | Percentage of Patients With Grade and Above Non-Hematologic Ti
Number analyzed (Participants) | 2
Participants
  Hypersensitivity Reaction | 1
  Fever | 1
  Nausea and Vomiting | 1
  Dehydration | 1

5. Primary Outcome: The Percentage of Patients Who Experience Any Grade of Peripheral Neuropathy
Description: The percentage of patients in the study who experience any grade of peripheral neuropathy during the study period
Time Frame: 583 days
Population: The two patients entered into the study were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Highly Sensitized Heart Transplant Candidates: Percentage of study patients with all grades of peripheral neuropathy during the study period
Arm/Group | Highly Sensitized Heart Transplant Candidates
Number analyzed (Participants) | 2
Participants | 1

6. Primary Outcome: Percentage of Patients Who Experience CMV, PTLD, and PML
Description: Percentage of patients who experience cytomegalovirus (CMV), post-transplant lymphoproliferative disease (PTLD), or progressive multifocal leukoencephalopathy (PML) during the study period.
Time Frame: 583 days
Population: The two patients who entered the study were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Incidnce of CMV, PTLD, PML: Percentage of patients who experience CMV, PTLD or PML within the study period
Arm/Group | Incidnce of CMV, PTLD, PML
Number analyzed (Participants) | 2
Participants | 0

7. Primary Outcome: The Percentage of Patients Who Experience Either a Respiratory Tract Infection or a Urinary Tract Infection
Description: The percentage of study patients who experience infectious complications in either the respiratory or urinary tracts during the study period.
Time Frame: 583 days
Population: The two patients who entered the study were evaluated
Measure: Count of Participants; unit: Participants
Groups:
- Respiratory Tract Infections: Number of Participants with Respiratory Tract Infections
- Urinary Tract Infections: Number of participants with urinary tract infections
Arm/Group | Respiratory Tract Infections | Urinary Tract Infections
Number analyzed (Participants) | 2 | 2
Participants | 1 | 1

8. Primary Outcome: The Percentage of Patients Who Experience Exacerbations Cardiac Dysrhythmias or Heart Failure
Description: The percentage of study patients who experience an exacerbation of cardiac dysrhythmias and heart failure during the study period
Time Frame: 583 days
Population: The two patients entered into the study were evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Patients With Exacerbation of Heart Failure: The study patients, who all have heart failure and need a heart transplant, but experience an exacerbation of their heart failure during the study period.
- Percentage of Patients With Exacerbation of Dysrythmias: The percentage of study patients who experienced an exacerbation of the incidence of cardiac dysrhythmias during the study period.
Arm/Group | Percentage of Patients With Exacerbation of Heart Failure | Percentage of Patients With Exacerbation of Dysrythmias
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

9. Primary Outcome: Percentage of Patients With Grade 4 Hematologic Toxicities
Description: A Grade 4 hematologic toxicity includes a platelet count < 25,000/mm3 or an absolute neutrophil count < 500/mm3
Time Frame: 583 days
Population: The two patient who entered the study were evaluated
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Patients With Grade 4 Hemotologic Toxicities: The percentage of patients who experienced a grade 4 hematologic toxicity as manifested by a platelet count < 25,000 mm3 or an absolute neutrophil count of < 500/mm3
Arm/Group | Percentage of Patients With Grade 4 Hemotologic Toxicities
Number analyzed (Participants) | 2
Participants | 0

10. Secondary Outcome: The Percentage of Patients With Antibody Mediated Rejection After Transplantation
Description: The percentage of patients who experience antibody mediated rejection at 6 months and 1 year post transplant. The study period was 583 days, during which a patient was eligible for transplant during the last 365 days. If a patient was transplanted on day 583, then the patient is followed for one year after the transplant, then the total time to assess the two patients would have been a period of two years or 730 days. In fact, neither patient was transplanted within the study period.
Time Frame: 730 days
Population: No study patient met the criteria for this measure since no patients were transplanted during the study period. The one patient who was eventually transplanted did not live to 6 months after the transplant.
Groups:
- Percentage of TX Patients With AMR at 6 Months: Percentage of study patients who were transplanted and then developed AMR by 6 months after transplant
- Percentage of TX Patients With AMR at 12 Months: The percentage of study patients who have developed AMR within 12 months of their transplant. This number includes those patients who had AMR diagnosed within 6 months of transplant.
Arm/Group | Percentage of TX Patients With AMR at 6 Months | Percentage of TX Patients With AMR at 12 Months
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Patients Who Develop De Novo Alloantibody or DSA Alloantibody After Transplant
Description: Percentage of patients who are transplanted with the study period who then develop de novo or donor-specific alloantibody (DSA) within one year post-transplant. The patients would be eligible for transplant after day 218 in the study protocol and the study had 365 days in which to be transplanted. If a patient was transplant on day 583,( the last day of eligibility), and then followed for one year, then the outcome time frame would be a total of two years. No patient was transplanted within the study period.
Time Frame: 730 days
Population: No patients met the criteria for this measure since the one patient eventually transplanted did not live long enough to develop donor specific antibodies.
Groups:
- Percentage of Pts. Who Develope De Novo or DSA < 1 yr After TX: Study patients who received a transplant and then developed de novo or donor specific antibodies after transplant.
Arm/Group | Percentage of Pts. Who Develope De Novo or DSA < 1 yr After TX
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Patients Post-Transplant That Are DSA Negative
Description: Percentage of patients who receive a transplant within the study period who are then DSA negative at 1 year following transplantation.
Time Frame: 730 days
Population: No patients were in this group
Groups:
- Percentage of Transplanted Pt That Are DSA Negative at 1 Year: Study patients who received a transplant during the study period and then are negative for donor specific antibodies at one year after transplant
Arm/Group | Percentage of Transplanted Pt That Are DSA Negative at 1 Year
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Allograft Survival
Description: The percentage of allografts transplanted during the study period that survive to 6 and 12 months post transplant.
Time Frame: 730 days
Population: No patients received a transplant during the study period. The one patient who was transplanted outside of the study period did not survive to 6 months.
Units Other Than Participants: Allografts
Groups:
- Allograft Survival at 6 Months: Study patients who receive a heart transplant within the study period whose allografts survive to 6 months.
- Allograft Survival at 12 Months: Study patients who are transplanted and whose allografts survive to one year. This number includes those allografts that survived to 6 months that then survived to 12 months.
Arm/Group | Allograft Survival at 6 Months | Allograft Survival at 12 Months
Number analyzed (Participants) | 0 | 0
Number analyzed (Allografts) | 0 | 0

14. Secondary Outcome: The Percentage of Allografts That Endure Acute Rejection Within One Year of Transplantation
Description: The percentage of allografts that have an acute rejection episode per the criteria of the International Society of Heart and Lung Transplantation (ISHLT) within one year of transplantation. Allografts implanted during the Recovery Phase are monitored for a year for acute rejection per the study protocol. An allograft potentially implanted on the last day of a patient's recovery period would still be monitored for a year, so the potential outcome measure time would be 730 days. Since no allografts were implanted during the recovery period, there are no results to report.
Time Frame: 730 days
Population: No patients met the criteria for this group. The one patient who received a transplant did not have the transplant during the study period, and she did not have signs of rejection at the time of her autopsy.
Groups:
- Percentage of Allografts With Acute Rejection: Allografts implanted within the study period are followed for one year after transplantation and are routinely monitored for allograft rejection.
Arm/Group | Percentage of Allografts With Acute Rejection
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Patients With a CPRA <20%, But Were Not Transplanted During the Study Period
Description: Proportion of patients who achieve a Calculated Panel Reactive Antibody test CPRA of < 20%, but are not transplanted within the study period.
Time Frame: 583 days
Population: No patients met this criteria since no patient had a CPRA of less than 20%.
Groups:
- Patients With CPRA < 20% Who Were Not Transplanted: Percentage of patients with a CPRA < 20% but not transplanted within one year
Arm/Group | Patients With CPRA < 20% Who Were Not Transplanted
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Patients Who Receive Transplants Who Then Suffer Serious Post-transplant Complications
Description: Percentage of study patients who receive transplants within the study period who then experience death, allograft loss, hospitalization due to infection, and non-fatal serious adverse cardiac event (defined as acute myocardial infarction, congestive heart failure, need for percutaneous cardiac intervention, coronary artery bypass grafting, cardiac defibrillator placement, cerebral vascular accident, peripheral vascular disease) within 1 year of transplantation.
Time Frame: 730 days
Population: No patients were transplanted within the study period so no patients could be analyzed for these potential outcomes
Groups:
- Transplant Patient Death: The incidence of death in transplanted patients at one year from transplant
- Allograft Loss in Transplanted Patients: Study patients who were transplanted and lost their allografts
- Hospitalization Due to Infection in Transplanted Patients: Study patients who were transplanted and then required hospitalization for infection within one year of the transplant
- Non-fatal Serious Cardiac Event: Study patients who were transplanted and had a non-fatal cardiac event(acute MI, congestive heart failure, coronary intervention, etc) at one year
Arm/Group | Transplant Patient Death | Allograft Loss in Transplanted Patients | Hospitalization Due to Infection in Transplanted Patients | Non-fatal Serious Cardiac Event
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from the initiation of study treatment through all three phases of the study the duration of which is 583 days. A patient could be transplanted on the last day of the recovery phase,(day 583), would then be followed for a year after the transplant for a total of 948 days
Groups:
- Study Treatment Group: All subjects will receive the study treatment. This is a non-randomized, open label study. The study treatment consists of an Induction phase with Thymoglobulin, Rituximab and Methylprednisolone, a Treatment phase with Bortezomib and a Recovery phase to follow-up and re-immunize and transplant the subject.
Arm/Group | Study Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Group (N=2)
Hospitalized with Hypersensitivity (Immune system disorders) | 1 (1) — Facial swelling, nausea and vomitting.
Hospitalized with Fever (General disorders) | 1 (1)
Hospitalized with LVAD Device Malfunction (Cardiac disorders) | 1 (2) — LVAD Device malfunction was device stopped.
Hospitalization for Nausea/Vomiting/Diarrhea (General disorders) | 1 (1)
Hospitalized with Dehydration (General disorders) | 1 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Group (N=2)
Bruising-Abdominal (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1) — Increased abdominal girth.
Pain-Abdominal (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2)
Pain-Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1)
Chest/Thorax NOS Pain (Cardiac disorders) | 1 (2) — Patient complained of chest pain during a device malfunction that resolved upon resolution of the malfunction.
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Decreased Bicarb (Investigations) | 1 (1) — Decreased Bicarb on study required lab work.
Decreased Hearing (Ear and labyrinth disorders) | 2 (3)
Decreased Hemoglobin (Investigations) | 2 (4) — Decreased Hemoglobin noted on study required lab work
Decreased Phosphate (Investigations) | 2 (2) — Decreased Phosphate on study required lab work.
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dizziness (Nervous system disorders) | 2 (4)
Dyspnes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated Uric Acid (Investigations) | 1 (1) — Elevated Uric Acid on study required lab work.
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 1 (1) — Elevated temperature with medication administration.
Headache (Nervous system disorders) | 1 (1)
Hot Flashes (Endocrine disorders) | 1 (1)
Hyperreaction to IVIG (Immune system disorders) | 2 (3)
Hypertension (Cardiac disorders) | 1 (1)
Hypocalcemia (Investigations) | 1 (1) — Decreased Calcium levels on study lab work.
Hypoglycemia (Investigations) | 1 (1) — Decreased Blood Glucose on study required lab work
Hypokalemia (Investigations) | 2 (4) — Decreased Potassium levels on study required lab work
Hypomagnesemia (Investigations) | 2 (5) — Decreased Magnesium levels on study required lab work.
Hypotension (Cardiac disorders) | 2 (6)
Incontinence (Renal and urinary disorders) | 2 (2)
Increased Creatinine (Investigations) | 1 (1) — Increased Creatinine on study required lab work.
Infection-Oral Cavity (Thrush) (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 1 (1)
Lower Extremity/Limb Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Foot cramping
Muscle cramps/pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (7)
Neuralgia/Peripheral Nerve Pain (Nervous system disorders) | 1 (1)
Neutropenia (Immune system disorders) | 1 (1)
Lower Extremity/Limb Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Leg Pain
Painful Urination (Renal and urinary disorders) | 1 (1)
Peripheral Edema (Blood and lymphatic system disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Serum Sickness (Immune system disorders) | 1 (1)
Stomach Ulcer (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Throat Pain (General disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Upper Extremity/Limb Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Shoulder Pain
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (6)
Ventricular Arrhythmias (Cardiac disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (4)
Difficulty Walking (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Weakness of left hand (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)
Bleeding from LVAD driveline site (Injury, poisoning and procedural complications) | 1 (1) — Pull on LVAD driveline that caused bleeding

LIMITATIONS AND CAVEATS:
The Study was terminated because of lack of efficacy. One patient was transplanted after the study period ended and died postoperatively. Autopsy did not reveal evidence of antibody mediated rejection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No